CLINICAL TRIAL: NCT03105349
Title: A Phase III, Open Label, Multicentric Clinical Trial of a Single Arm of 16 Weeks of Duration to Evaluate Retreatment With Elbasvir/Grazoprevir Plus Sofosbuvir and Ribavirin in Patients With Chronic Hepatitis C Genotype 1,4 Who Have Failed to Treat With a Regime Based on an Inhibitor of the NS5A
Brief Title: A Clinical Trial of 16 Weeks of Duration to Evaluate Retreatment With Elbasvir/Grazoprevir Plus Sofosbuvir and Ribavirin in Patients With Chronic Hepatitis C Genotypes 1,4 Who Have Failed to Treat With a Regime Based on an Inhibitor of the NS5A
Acronym: C-RESCUE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No availability of investigational medication.
Sponsor: Fundacion SEIMC-GESIDA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA 9516
Record Dates: First submitted 2017-03-16; First posted 2017-04-07 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: HCV
MeSH Terms: interventions — elbasvir-grazoprevir drug combination; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): 16 weeks treatment with elbasvir/grazoprevir plus sofosbuvir and ribavirina
  Interventions: Drug: elbasvir/grazoprevir; Drug: Sofosbuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: elbasvir/grazoprevir — 16 weeks treatment
  Other Names: Zepatier
Drug: Sofosbuvir — 16 weeks treatment
Drug: Ribavirin — 16 weeks treatment

SUMMARY:
This is a phase 4 clinical trial to treat patients who have failed to treat with regimen based on an inhibitor of the NS5A

DETAILED DESCRIPTION:
The duration of the treatment will be 16 weeks and then will be a security perid with 2 visits (Week 12 post treatment and week 24 post treatment) The study in an open label study with a single arm .

ELIGIBILITY:
Inclusion Criteria:

* Adults with chronic HCV genotype 1, 4 infection with or without HIV infection aged 18 years or above
* HCV RNA plasma concentration of at least 1000 IU / mL
* Subjects previously treated with NS5A-based regimens for at least 8 weeks.
* Patients with HCV relapse after receiving a complete treatment with NS5A-based AAD regimen for at least 8 weeks and becoming undetectable at the end of treatment. Relapse is defined as a confirmed HCV RNA detectable upon completion of therapy of A5 based on NS5A against HCV.
* Subjects with compensated hepatic cirrhosis (Child A) could be included.
* For patients with HIV coinfection:

  * Be infected with HIV-1, documented by any rapid HIV test with the corresponding license and confirmed by a Western blot or second antibody test using a method other than the initial rapid HIV and / or I / CIA method or by HIV-1 p24 antigen or viral load of HIV-1 RNA plasma.
  * Be on stable HIV antiretroviral therapy (ART) for at least 4 weeks prior to entry into the study using a dual ITN backbone of tenofovir or abacavir and emtricitabine or lamivudine PLUS raltegravir or dolutegravir or rilpivirine (with CD4 + T cell count> 100 cells / mm 3 and undetectable HIV-1 RNA at baseline. Results from prior analysis will be accepted within 24 weeks prior to study entry).

Exclusion Criteria:

* Subjects with hepatitis other than C or steatosis.
* Subjects previously treated less than 8 weeks with regimens based on NS5A.
* Evidence of previous hepatocellular carcinoma although it has criteria of cure
* Subjects with past or current decompensated liver disease; Only decompensated patients who have received a liver transplant and have not decompensated after transplantation will be included.
* Subjects suspected of clinical or genotypic reinfection of HCV.
* Subject with HCV response regrowth while receiving NS5A-based ADA therapy against HCV. Said regrowth is defined as a confirmation of detectable HCV RNA after achieving undetectable HCV RNA during NS5A-based AADs against HCV.
* Recent history of drug or alcohol abuse.
* Important comorbidities.

  * Pregnant, lactating or non-lactating women Contraceptives, if they are women of childbearing age. Women of childbearing age are defined as those women who have not undergone permanent infertility procedures or who have been amenorrheic for less than 12 months.
  * Subjects with a glomerular filtration rate of less than 30 ml / min.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
The rate of patients achieved SVR12 | Week 12 post treatment

SECONDARY OUTCOMES:
The proportion of subjects infected with HCV genotype 1a with reference VARs NS5A / NS3 who achieved RVS12. | Week 12 post treatment
  To analyze the impact of VARs NS5A/NS3 on RVS12
The proportion of subjects infected with HCV genotype 1b with reference VARs NS5A / NS3 who achieved RVS12. | Week 12 post treatment
  Analyze the impact of VARs NS5A/NS3 on RVS12
The proportion of subjects infected with HCV genotype 4 with reference VARs NS5A /NS3 who achieved RVS12. | Week 12 post treatment
  Analyze the impact of VARs NS5A/NS3 on RVS12
The proportion of subjects infected with HCV genotypes 1.4 with reference VARs NS5A /NS3 who achieved RVS24. | Week 24 post treatment
  Analyze the impact of VARs NS5A/NS3 on RVS24
The occurrence of Viral resistance variants (VARs) to NS5A or elbasvir, to NS3 or grazoprevir and to NS5B or SOF in patients who did not reach SVR12 after 16 weeks of re-treatment | Week 16
  the occurrence of resistance in patients who did not reach SVR12 after 16 weeks of re-treatment
The occurrence of resistance variants (VARs) viral to NS5A or elbasvir, to NS3 or grazoprevir, and to NS5B or SOF in HIV patients included | Week 12 post treatment
  The impact of VARs NS5A/NS3 on RVS12
  The proportion of subjects developing HIV-1 virological failure (HIV RNA> 200 Copies / mL), confirmed in 2 consecutive tests with at least 2 weeks between them.
The proportion of subjects developing HIV-1 virological failure (HIV RNA> 200 Copies / mL), confirmed in 2 consecutive tests with at least 2 weeks between them | Week 4, week 8, week 12 and week 16
  the impact of treatment with EL / BRA plus SOFT and ribavirin in HIV-1 subjects
The proportion of subjects experiencing adverse events of high laboratory values who report as ECI at any time during the study period. | Week 4, week 8, week 12, week 16, week 12 post-treatment and week 24 post-treatment
  Adverse events
The proportion of subjects with at least one adverse experience | Week 4, week 8, week 12, week 16, week 12 post-treatment and week 24 post-treatment
  Adverse events
The proportion of subjects with an adverse experience related to medication | Week 4, week 8, week 12, week 16, week 12 post-treatment and week 24 post-treatment
  Adverse events
The proportion of subjects with a severe adverse experience | Week 4, week 8, week 12, week 16, week 12 post-treatment and week 24 post-treatment
  Adverse events
The proportion of subjects with a serious adverse experience related to medication | Week 4, week 8, week 12, week 16, week 12 post-treatment and week 24 post-treatment
  Adverse events
The proportion of subjects with an adverse experience leading to disruption | Week 4, week 8, week 12, week 16, week 12 post-treatment and week 24 post-treatment
  Adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Univ. La Paz, Madrid, Madri
  - Hospital Univ. Gregorio Marañon, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospita 12 de octubre, Madrid
  - Hospital Univ. La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No